CLINICAL TRIAL: NCT05494736
Title: A Single-Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics, and Anti-Retroviral Activity of MK-8527 Monotherapy in Anti-Retroviral Therapy (ART)-Naïve, HIV-1 Infected Participants
Brief Title: MK-8527 Single-Dose Trial in HIV-1 Infected Participants (MK-8527-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8527-004; MK-8527-004 (Other: Merck); 2023-503682-39 (Registry Identifier: EU CT); U1111-1287-7295 (Registry Identifier: UTN)
Record Dates: First submitted 2022-08-02; First posted 2022-08-10 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Panel A: MK-8527 1.0 mg (Experimental): Participants receive a single oral dose of MK-8527 1.0 mg.
  Interventions: Drug: MK-8527
- Panel B: MK-8527 0.5 mg (Experimental): Participants receive a single oral dose of MK-8527 0.5 mg.
  Interventions: Drug: MK-8527
- Panel C: MK-8527 0.25 mg (Experimental): Participants receive a single oral dose of MK-8527 0.25 mg.
  Interventions: Drug: MK-8527

INTERVENTIONS:
Drug: MK-8527 — MK-8527 capsule taken by mouth.

SUMMARY:
This is a single-dose clinical study to evaluate the safety, tolerability, pharmacokinetics, and anti-retroviral activity of MK-8527 in antiretroviral therapy (ART)-naïve participants living with human immunodeficiency virus type 1 (HIV-1) infection. The primary hypothesis is that, at a dose that is safe and generally well tolerated, MK-8527 will have antiretroviral activity as measured by a reduction from baseline in plasma HIV-1 ribonucleic acid (RNA) of ≥1.0 log10 copies/mL. A total of 4 arms was initially planned but Arm D was never initiated as the primary objectives were achieved following completion of Arms A to C.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health other than HIV-1 infection
* Is documented HIV-1 positive
* Is ART-naïve, which is defined as not having received any marketed antiretroviral agent for treatment of HIV-1 infection (prior use of an ART for PrEP or investigational therapy is permitted if the last dose was ≥30 days prior to study drug administration)
* Is willing to receive no other ART for the monitoring period of this study

Exclusion Criteria:

* Has a history of clinically significant endocrine, GI, cardiovascular, hematological, hepatic, immunological (outside of HIV-1 infection), renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study intervention, throughout the study, until the poststudy visit
* Has participated in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to the prestudy (screening) visit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- ARENSIA Exploratory Medicine-Institutul National de Boli Infectioase Matei Bals ( Site 0004), Bucharest, București, Romania
- South Africa (3):
  - Josha Research ( Site 0003), Bloemfontein, Free State
  - Helen Joseph Hospital-Clinical HIV Research Unit ( Site 0002), Johannesburg, Gauteng
  - Desmond Tutu Health Foundation ( Site 0001), Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26180&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were recruited at study sites in Romania and South Africa. A total of 4 arms was initially planned, but Arm D was never initiated as the primary objectives were achieved following completion of Arms A to C.
Groups:
- Panel A: MK-8527 1.0 mg: Participants receive a single oral dose of MK-8527 1.0 mg on Day 1.
- Panel B: MK-8527 0.5 mg: Participants receive a single oral dose of MK-8527 0.5 mg on Day 1.
- Panel C: MK-8527 0.25 mg: Participants receive a single oral dose of MK-8527 0.25 mg on Day 1.
Period: Overall Study
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Started | 8 | 6 | 6
Completed | 8 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were no participants in Panel D.
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (8.6) | 23.8 (3.5) | 37.8 (12.6) | 30.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 2 | 13
  Male | 3 | 0 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 6 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 6 | 2 | 16
  White | 0 | 0 | 4 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma HIV-1 Ribonucleic Acid (RNA)
Description: The mean change from baseline in HIV-1 RNA counts at 168 hours after a single doses of MK-8527 is reported.
Time Frame: Baseline and 168 hours postdose on Day 1
Population: All participants who complied with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model, are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: HIV-1 RNA copies/mL
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 6
HIV-1 RNA copies/mL | -1.38 [-1.61 to -1.15] | -1.40 [-1.66 to -1.13] | -0.80 [-1.06 to -0.53]

2. Primary Outcome: Number of Participants Experiencing ≥1 Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 28 days
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 6
Participants | 5 | 5 | 2

3. Primary Outcome: Number of Participants Discontinuing From Study Due to an AE
Description: as for outcome 2
Time Frame: Up to 28 days
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 6
Participants | 0 | 0 | 0

4. Secondary Outcome: Area Under the Concentration-Time Curve From Predose to 168 Hours Postdose (AUC0-168) of MK-8527 Triphosphate (MK-8527-TP) in Peripheral Blood Mononuclear Cells (PBMCs)
Description: The AUC0-168 of MK-8527-TP in PBMCs is reported.
Time Frame: Predose and 4, 12, 24, 96, 120, 144, and 168 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: h*pmol/10^6 cells
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 6
h*pmol/10^6 cells | 29.2 [24.1 to 35.3] | 12.6 [10.1 to 15.7] | 5.53 [4.44 to 6.89]

5. Secondary Outcome: Area Under the Concentration-Time Curve From Predose to Infinity (AUC0-inf) of MK-8527-TP in PBMCs
Description: The MK-8527-TP AUC0-inf in PBMCs is reported.
Time Frame: Predose and 4, 12, 24, 96, 120, 144, 168, 192, 240, 336, 504, and 672 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: h*pmol/10^6 cells
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 5
h*pmol/10^6 cells | 47.7 [37.8 to 60.3] | 24.5 [18.7 to 32.1] | 8.87 [6.60 to 11.9]

6. Secondary Outcome: Area Under the Concentration-Time Curve From Predose to Last Measurable Concentration (AUC0-last) of MK-8527-TP in PBMCs
Description: The MK-8527-TP AUC0-last in PBMCs is reported.
Time Frame: Predose and 4, 12, 24, 96, 120, 144, 168, 192, 240, 336, 504, and 672 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: h*pmol/10^6 cells
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 6
h*pmol/10^6 cells | 40.9 [32.5 to 51.4] | 17.1 [13.1 to 22.2] | 5.88 [4.51 to 7.66]

7. Secondary Outcome: Maximum Concentration (Cmax) of MK-8527-TP in PBMCs
Description: The MK-8527-TP Cmax in PBMCs is reported.
Time Frame: Predose and 4, 12, 24, 96, 120, 144, 168, 192, 240, 336, 504, and 672 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/10^6 cells
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 6
pmol/10^6 cells | 0.270 [0.232 to 0.314] | 0.134 [0.113 to 0.160] | 0.0535 [0.0449 to 0.0637]

8. Secondary Outcome: Concentration at 168 Hours Postdose (C168) of MK-8527-TP in PBMCs
Description: The C168 of MK-8527-TP in PBMCs is reported.
Time Frame: 168 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/10^6 cells
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 7 | 6 | 6
pmol/10^6 cells | 0.111 [0.0808 to 0.152] | 0.0484 [0.0344 to 0.0681] | 0.0224 [0.0154 to 0.0325]

9. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-8527-TP in PBMCs
Description: The MK-8527-TP Tmax in PBMCs is reported.
Time Frame: Predose and 4, 12, 24, 96, 120, 144, 168, 192, 240, 336, 504, and 672 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 6
hours | 24.00 [12.00 to 24.05] | 24.03 [12.07 to 24.68] | 23.91 [12.00 to 24.12]

10. Secondary Outcome: Apparent Terminal Half-life (t½) of MK-8527-TP in PBMCs
Description: The apparent t½ of MK-8527-TP in PBMCs is reported.
Time Frame: Predose and 4, 12, 24, 96, 120, 144, 168, 192, 240, 336, 504, and 672 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 5
Hours | 128.24 (49.00) | 172.09 (90.23) | 80.15 (52.35)

11. Secondary Outcome: AUC0-inf of MK-8527 in Plasma
Description: The AUC0-inf of MK-8527 in plasma is reported.
Time Frame: Predose and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours postdose
Population: All participants who complied with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model, are included. Participants with data below the lower limit of quantification (LLOQ) are excluded.
Measure: Geometric Mean (95% Confidence Interval); unit: h*umol/L
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 7 | 6 | 6
h*umol/L | 0.0512 [0.0360 to 0.0728] | NA [NA to NA] — For all the participants in Panel B and Panel C, only 1 or 2 concentration samples were measurable (in the absorption phase) out of 11 sampling time points collected. All the other concentration data were BLOQ. Therefore, the plasma PK parameters requiring measurable concentrations in the terminal phase were not evaluated for the participants in Panel B and Panel C. | NA [NA to NA] — For all the participants in Panel B and Panel C, only 1 or 2 concentration samples were measurable (in the absorption phase) out of 11 sampling time points collected. All the other concentration data were BLOQ. Therefore, the plasma PK parameters requiring measurable concentrations in the terminal phase were not evaluated for the participants in Panel B and Panel C.

12. Secondary Outcome: AUC0-last of MK-8527 in Plasma
Description: The AUC0-last of MK-8527 in plasma is reported.
Time Frame: Predose and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours postdose
Population: All participants who complied with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model, are included.
  Participants with data below the LLOQ are excluded.
Measure: Geometric Mean (95% Confidence Interval); unit: h*umol/L
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 6
h*umol/L | 0.0304 [0.0221 to 0.0419] | NA [NA to NA] — For all the participants in Panel B and Panel C, only 1 or 2 concentration samples were measurable (in the absorption phase) out of 11 sampling time points collected. All the other concentration data were BLOQ. Therefore, the plasma PK parameters requiring measurable concentrations in the terminal phase were not evaluated for the participants in Panel B and Panel C. | NA [NA to NA] — For all the participants in Panel B and Panel C, only 1 or 2 concentration samples were measurable (in the absorption phase) out of 11 sampling time points collected. All the other concentration data were BLOQ. Therefore, the plasma PK parameters requiring measurable concentrations in the terminal phase were not evaluated for the participants in Panel B and Panel C.

13. Secondary Outcome: Clast of MK-8527 in Plasma
Description: The Clast of MK-8527 in plasma is reported.
Time Frame: Predose and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours postdose
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 5
umol/L | 0.00388 [0.00346 to 0.00435] | 0.00433 [0.00380 to 0.00495] | 0.00417 [0.00361 to 0.00482]

14. Secondary Outcome: Cmax of MK-8527 in Plasma
Description: The Cmax of MK-8527 in plasma is reported.
Time Frame: Predose and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours postdose
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 5
umol/L | 0.0224 [0.0172 to 0.0292] | 0.00935 [0.00688 to 0.0127] | 0.00469 [0.00335 to 0.00656]

15. Secondary Outcome: Tmax of MK-8527 in Plasma
Description: The Tmax of MK-8527 in plasma is reported.
Time Frame: Predose and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours postdose
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 8 | 6 | 5
Hours | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 3.00] | 0.50 [0.23 to 1.00]

16. Secondary Outcome: Apparent t½ of MK-8527 in Plasma
Description: The apparent t½ of MK-8527 in plasma is reported.
Time Frame: Predose and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours postdose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg
Number analyzed (Participants) | 7 | 6 | 6
Hours | 3.25 (54.52) | NA (NA) — For all the participants in Panel B and Panel C, only 1 or 2 concentration samples were measurable (in the absorption phase) out of 11 sampling time points collected. All the other concentration data were BLOQ. Therefore, the plasma PK parameters requiring measurable concentrations in the terminal phase were not evaluated for the participants in Panel B and Panel C. | NA (NA) — For all the participants in Panel B and Panel C, only 1 or 2 concentration samples were measurable (in the absorption phase) out of 11 sampling time points collected. All the other concentration data were BLOQ. Therefore, the plasma PK parameters requiring measurable concentrations in the terminal phase were not evaluated for the participants in Panel B and Panel C.

17. Secondary Outcome: Correlation Between Intracellular C168 of MK-8527-TP in PBMCs and Change From Baseline in Plasma HIV-1 RNA
Description: The correlation between between the C168 of MK-8527-TP in PBMCs and the change from baseline in plasma HIV-1 RNA levels 168 hours after dosing was calculated based on all pooled participants. All participants who complied with the protocol sufficiently to ensure that generated data will belikely to exhibit the effects of treatment, according to the underlying scientific model, are included. Participants with data below the LLOQ are excluded.
Time Frame: Predose and 168 hours postdose
Population: as for outcome 1
Measure: Number; unit: Pearson r coefficient
Groups:
- Panels A to C: MK-8527 Pooled: All participants who received a single oral dose of MK-8527 are included.
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel C: MK-8527 0.25 mg | Panels A to C: MK-8527 Pooled
Number analyzed (Participants) | 8 | 6 | 6 | 20
Pearson r coefficient | NA — All arms were pooled to calculate Pearson r. | NA — All arms were pooled to calculate Pearson r. | NA — All arms were pooled to calculate Pearson r. | -0.342

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: All participants who received ≥1 dose of study drug are included.
Groups:
- Panel D: MK-8527 0.25 mg: Participants receive a single oral dose of MK-8527 0.25 mg on Day 1.
Arm/Group | Panel A: MK-8527 1.0 mg | Panel B: MK-8527 0.5 mg | Panel D: MK-8527 0.25 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/8 | 5/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panel A: MK-8527 1.0 mg (N=8) | Panel B: MK-8527 0.5 mg (N=6) | Panel D: MK-8527 0.25 mg (N=6)
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vessel puncture site bruise (General disorders) | 0 | 1 | 0
Impetigo (Infections and infestations) | 1 | 1 | 0
Tinea faciei (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Carbuncle (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Viral rash (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT05494736/Prot_SAP_000.pdf